CLINICAL TRIAL: NCT00909935
Title: The Pharmacokinetics of Dexmedetomidine in Children
Status: Terminated | Type: Observational
Why Stopped: unable to enroll enough patients
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Keira Mason, Senior Associate in Perioperative Anesthesia, Boston Children's Hospital
Other Study IDs: 09-02-0067
Record Dates: First submitted 2009-04-30; First posted 2009-05-29 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: MRI Sedation
Keywords: To determine pharmacokinetics of dexmedetomidine in children
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Dexmedetomidine — Initial 2 mcg/kg bolus administered over 10 minutes to achieve the Ramsey sedation score of 4 followed by an infusion of 1.5 mcg/kg/hr, which will run until patient is transferred to recovery area. Up to a further two boluses of 2 mcg/kg may be given to maintain an RSS of 4.
  Other Names: Precedex

SUMMARY:
This study is designed to identify the plasma concentrations which are required to achieve adequate sedation, using a Ramsay Sedation Scale. As an alpha 2 agonist, dexmedetomidine can elicit hemodynamic changes, fluctuations in blood pressure and heart rate. This study will attempt to determine whether these changes can be predicted by plasma concentrations.

DETAILED DESCRIPTION:
Dexmedetomidine, an alpha2 agonist is currently the standard of care for sedation for diagnostic (MRI, CT and Nuclear Medicine) radiological studies at Boston Children's Hospital. Although it is FDA approved for sedation, its pharmacokinetics in children has not been carefully studied with prospective studies. The plasma concentration of dexmedetomidine necessary to achieve and maintain adequate sedation for motionless conditions for a MRI study has not been determined which is the purpose of this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 - 11.9 years

  * 2 age groups: 3.0 - 5.9 years, 6.0 - 11.9 years
* Patients will be equally distributed within each age group
* Meets criteria to receive dexmedetomidine sedation for MRI:

  * Active, uncontrolled gastroesophageal reflux - an aspiration risk
  * Active, uncontrolled vomiting - an aspiration risk
  * Current (or within past 3 months) history of apnea requiring an apnea monitor
  * Active, current respiratory issues that are different from the baseline status (pneumonia,exacerbation of asthma, bronchiolitis, respiratory syncytial virus)
  * Unstable cardiac status (life threatening arrhythmias, abnormal cardiac anatomy,significant cardiac dysfunction)
  * Craniofacial anomaly, which could make it difficult to effectively establish a mask airway for positive pressure ventilation if needed
  * Current use of digoxin
  * Moya Moya Disease
  * New-onset stroke
  * Provide written consent to take part in the research study

Exclusion Criteria:

* Do not meet established sedation criteria
* History of allergy, intolerance, or reaction to dexmedetomidine or hypersensitivity
* Previous diagnosis of hepatic insufficiency/failure or a serum glutamate pyruvate transaminase level > 2 times the normal limit determined by Children's Hospital Boston (TCH)
* Current diagnosis of renal insufficiency/failure or a current serum creatinine level > 1.5 times the normal limit determined by TCH
* Have received digoxin in the past (no time limit)
* Received phenobarbital, clonidine or valproic acid within 30 days
* Current, repaired or risk of Moya-Moya disease
* Recent stroke (cerebrovascular accident) within past 6 months
* Uncontrolled hypertension
* Concomitant use of beta antagonist, or calcium channel blocker
* Participated in a clinical investigation within the past three months

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children requiring sedation for MRI scanning
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of dexmedetomidine in pediatric patients | 2012-2015

CONTACTS AND LOCATIONS:
Overall Officials: Keira P. Mason, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States